CLINICAL TRIAL: NCT07319182
Title: Accuracy of Artificial Intelligence Technology in Detecting Periapical Lesions in Human Teeth. Diagnostic Accuracy Experimental Study.
Brief Title: Accuracy of Artificial Intelligence Technology in Detecting Periapical Lesions in Human Teeth.
Acronym: AI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Mays Maher Albochi, Master Student, Future University in Egypt
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: (52)/11-2024
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Periapical Lesion
Keywords: artificial intelligence, periapical lesion, CBCT

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cone beam computed tomography (Active Comparator): detecting radiolucent periapical lesions using cone beam computed tomography
  Interventions: Other: Cone beam computed tomography
- artificial intelligence software (Active Comparator): Cone beam CT scan will be uploaded to artificial intelligence software to ensure that the software will detect radiolucent periapical lesion compared to Cone beam CT scans.
  Interventions: Other: artificial intelligence software

INTERVENTIONS:
Other: Cone beam computed tomography — Cone beam computed tomography scans to detect the presence of periapical lesion by specialized investigators.
  Arms: cone beam computed tomography
Other: artificial intelligence software — artificial intelligence software that aids in diagnosis in dentistry
  Arms: artificial intelligence software

SUMMARY:
Aims to evaluate the accuracy of using Artificial intelligence software in detecting the presence of periapical lesion compared to CBCT imaging.

DETAILED DESCRIPTION:
In this research, patients referred to endodontic department in the university will undergo clinical examination (percussion, palpation) tests. These will be recorded. Then the patient will undergo a periapical radiograph to detect the presence of periapical lesion. Patients with periapical lesions will then undergo a cone beam computed tomography and this scan will be uploaded into the Artificial intelligence software to detect the accuracy of the software in detecting the presence of the periapical lesion. Any patient with a periapical lesion in need of root canal treatment will undergo the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be medically free from any systemic disease that can affect root canal treatment.
2. 18 to 50 years old patients with permanent teeth presenting with periapical pathosis.
3. No sex predilection.
4. All patients must have good oral hygiene.
5. Restorable teeth
6. Positive patient's acceptance for participating in the study.
7. Patients able to sign informed consent

Exclusion Criteria:

1. Patients above 50 years or patients below 18 years.
2. Patients with very poor oral hygiene.
3. Pregnant women after taking detailed history and pregnancy test must be in the first visit.
4. Psychologically disturbed patients.

Teeth that have:

* Periodontally affected with grade 2 or 3 mobility.
* Not restorable teeth.
* Abnormal anatomy and calcified canals

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-21 (Actual)

PRIMARY OUTCOMES:
CBCT scans | 1 year
  Presence of periapical lesion on CBCT scans

SECONDARY OUTCOMES:
Accuracy of Artificial intelligence software | 1 year
  Comparing results from CBCT scans to Artificial intelligence software in detection of periapcial lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Future University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: within 1 year from registering the study protocol
Access Criteria: within 1 year from registering the study protocol